CLINICAL TRIAL: NCT02343016
Title: Evaluation of NIRS as a Continuous Noninvasive Monitoring System of Liver/Kidney Graft Perfusion in the Early Postoperative Period in Pediatric Patients. Pilot Study
Brief Title: NIRS as a Continuous Noninvasive Monitoring System of Liver/Kidney Graft Perfusion
Acronym: NIRS
Status: Terminated | Type: Observational
Why Stopped: due to a decision by the research team not to continuos the study
Sponsor: Mariella Enoc (Other)
Collaborators: Medtronic - MITG (Industry)
Responsible Party: Sponsor-Investigator, Mariella Enoc, Dirigente Medico A.R.C.O., Bambino Gesù Hospital and Research Institute
Organization: Bambino Gesù Hospital and Research Institute (Other)
Other Study IDs: 781_OPBG_2014
Record Dates: First submitted 2014-11-10; First posted 2015-01-21 (Estimated); Last update posted 2019-05-22 (Actual); Status verified 2019-05

CONDITIONS: Liver Failure; Kidney Failure
MeSH Terms: conditions — Liver Failure; Renal Insufficiency | interventions — Spectroscopy, Near-Infrared

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — * Blood count
  * Coagulation: INR, PT,PTT, ATIII, fibrinogen
  * Electrolytes
  * Albumine, proteins
  * Liver function specific markers: GOT/GPT, total and direct bilirubin, urea nitrogen, lactic acid
  * Renal function specific markers: NGAL, creatinine, urea nitrogen
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Near-InfraRed Spectroscopy (NIRS): The NIRS Group will be monitored with the interventional system (NIRS) and with the standard one (ecodoppler)
  Interventions: Device: Near-InfraRed Spectroscopy (NIRS)

INTERVENTIONS:
Device: Near-InfraRed Spectroscopy (NIRS) — NIRS is a non invasive monitoring system that enables assessment of tissue oxygenation through a quantitative estimation of haemoglobin oxygen-saturation within tissues.
  Other Names: Somanetics INVOS® system

SUMMARY:
The aim of the investigators work is to describe the agreement between NIRS and ecodoppler, as monitoring systems of liver and kidney graft's perfusion in the immediate postoperative period in pediatric patients.

DETAILED DESCRIPTION:
This is an observational descriptive pilot study to explore the Somanetics INVOS® system performance. In this study the investigators will recruit a convenient number of patients, 15 patients, that will be admitted to our ICU after liver/kidney transplantation, in a 6 month period.

The Primary endpoint will be the correlation between hepatic/renal NIRS measurements and graft's artery resistance indices, as evaluated with ecodoppler.

The Secondary endpoints will be:

* The Correlation between NIRS measurements and biochemical indicators of graft function (NGAL for kidney transplantation and INR, SGOT/SGPT, bilirubin, lactate for liver transplantation)
* The Correlation between NIRS measurements and SvO2 values

ELIGIBILITY:
Inclusion Criteria:

* All pediatric patients admitted to our ICU for postoperative care after liver/kidney transplantation

Exclusion Criteria:

* Obesity (BMI > 35)
* Presence of a surgical plate over the graft
* Impossibility of probe positioning, because of surgical wound, medication or drainage
* Bilirubin level > 30 mg/dL

Max Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: All pediatric patients admitted to our ICU for postoperative care after liver/kidney transplantation.
Sampling Method: Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2015-02 (Actual); Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
hepatic/renal NIRS measurements and graft's artery resistance indices, as evaluated with ecodoppler | every hour from recovery time to 6 hours after extubation

SECONDARY OUTCOMES:
hepatic/renal NIRS measurements and biochemical indicators of graft function: - NGAL for kidney transplantation - INR, SGOT/SGPT, bilirubin, lactate for liver transplantation | every hour until from recovery to 6 hours after extubation
hepatic/renal NIRS measurements and SvO2 values | every hour from recovery to 6 hours after extubation

CONTACTS AND LOCATIONS:
Overall Officials: Sergio Picardo, MD, Study Director — Bambino Gesù Hospital and Research Institute
Locations (1):
- Bambino Gesù Hospital and Research Institute, Rome, Italy

REFERENCES:
- [Background] Spada M, Riva S, Maggiore G, Cintorino D, Gridelli B. Pediatric liver transplantation. World J Gastroenterol. 2009 Feb 14;15(6):648-74. doi: 10.3748/wjg.15.648. PMID 19222089
- [Background] Hendrickson RJ, Karrer FM, Wachs ME, Slater K, Bak TE, Kam I. Pediatric liver transplantation. Curr Opin Pediatr. 2004 Jun;16(3):309-13. doi: 10.1097/01.mop.0000127160.82531.77. PMID 15167019
- [Background] Ghobrial RM, Farmer DG, Amersi F, Busuttil RW. Advances in pediatric liver and intestinal transplantation. Am J Surg. 2000 Nov;180(5):328-34. doi: 10.1016/s0002-9610(00)00550-x. PMID 11137682
- [Background] Jobsis FF. Noninvasive, infrared monitoring of cerebral and myocardial oxygen sufficiency and circulatory parameters. Science. 1977 Dec 23;198(4323):1264-7. doi: 10.1126/science.929199.
- [Background] Mancini DM, Bolinger L, Li H, Kendrick K, Chance B, Wilson JR. Validation of near-infrared spectroscopy in humans. J Appl Physiol (1985). 1994 Dec;77(6):2740-7. doi: 10.1152/jappl.1994.77.6.2740. PMID 7896615
- [Background] Ghanayem NS, Wernovsky G, Hoffman GM. Near-infrared spectroscopy as a hemodynamic monitor in critical illness. Pediatr Crit Care Med. 2011 Jul;12(4 Suppl):S27-32. doi: 10.1097/PCC.0b013e318221173a. PMID 22129547
- [Background] Beilman GJ, Groehler KE, Lazaron V, Ortner JP. Near-infrared spectroscopy measurement of regional tissue oxyhemoglobin saturation during hemorrhagic shock. Shock. 1999 Sep;12(3):196-200. doi: 10.1097/00024382-199909000-00005. PMID 10485597
- [Background] Moerman A, Wouters P. Near-infrared spectroscopy (NIRS) monitoring in contemporary anesthesia and critical care. Acta Anaesthesiol Belg. 2010;61(4):185-94. PMID 21388077
- [Background] Johnson BA, Chang AC. Near-infrared spectroscopy and tissue oxygenation: the unremitting quest for the holy grail. Pediatr Crit Care Med. 2008 Jan;9(1):123-4. doi: 10.1097/01.PCC.0000299375.17007.BC. No abstract available. PMID 18185128
- [Background] Nagdyman N, Fleck T, Schubert S, Ewert P, Peters B, Lange PE, Abdul-Khaliq H. Comparison between cerebral tissue oxygenation index measured by near-infrared spectroscopy and venous jugular bulb saturation in children. Intensive Care Med. 2005 Jun;31(6):846-50. doi: 10.1007/s00134-005-2618-0. Epub 2005 Apr 1. PMID 15803294
- [Background] Nagdyman N, Ewert P, Peters B, Miera O, Fleck T, Berger F. Comparison of different near-infrared spectroscopic cerebral oxygenation indices with central venous and jugular venous oxygenation saturation in children. Paediatr Anaesth. 2008 Feb;18(2):160-6. doi: 10.1111/j.1460-9592.2007.02365.x. PMID 18184248
- [Background] El-Desoky AE, Jiao LR, Havlik R, Habib N, Davidson BR, Seifalian AM. Measurement of hepatic tissue hypoxia using near infrared spectroscopy: comparison with hepatic vein oxygen partial pressure. Eur Surg Res. 2000;32(4):207-14. doi: 10.1159/000008766. PMID 11014921
- [Background] Mitsuta H, Ohdan H, Fudaba Y, Irei T, Tashiro H, Itamoto T, Asahara T. Near-infrared spectroscopic analysis of hemodynamics and mitochondrial redox in right lobe grafts in living-donor liver transplantation. Am J Transplant. 2006 Apr;6(4):797-805. doi: 10.1111/j.1600-6143.2006.01247.x. PMID 16539638
- [Background] Fortune PM, Wagstaff M, Petros AJ. Cerebro-splanchnic oxygenation ratio (CSOR) using near infrared spectroscopy may be able to predict splanchnic ischaemia in neonates. Intensive Care Med. 2001 Aug;27(8):1401-7. doi: 10.1007/s001340100994. PMID 11511955
- [Background] Leone M, Blidi S, Antonini F, Meyssignac B, Bordon S, Garcin F, Charvet A, Blasco V, Albanese J, Martin C. Oxygen tissue saturation is lower in nonsurvivors than in survivors after early resuscitation of septic shock. Anesthesiology. 2009 Aug;111(2):366-71. doi: 10.1097/ALN.0b013e3181aae72d. PMID 19602965
- [Background] Mulier KE, Skarda DE, Taylor JH, Myers DE, McGraw MK, Gallea BL, Beilman GJ. Near-infrared spectroscopy in patients with severe sepsis: correlation with invasive hemodynamic measurements. Surg Infect (Larchmt). 2008 Oct;9(5):515-9. doi: 10.1089/sur.2007.091. PMID 18687043
- [Background] Nanas S, Gerovasili V, Renieris P, Angelopoulos E, Poriazi M, Kritikos K, Siafaka A, Baraboutis I, Zervakis D, Markaki V, Routsi C, Roussos C. Non-invasive assessment of the microcirculation in critically ill patients. Anaesth Intensive Care. 2009 Sep;37(5):733-9. doi: 10.1177/0310057X0903700516. PMID 19775036